CLINICAL TRIAL: NCT05891899
Title: Antithrombin Registry - Investigation of Phenotype-genotype Correlations in Patients With Inherited Antithrombin Deficiency
Brief Title: Belgian Antithrombin Deficiency Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Christelle Orlando, Professor, Universitair Ziekenhuis Brussel
Other Study IDs: UZB-ATRegistry
Record Dates: First submitted 2023-05-12; First posted 2023-06-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Antithrombin III Deficiency
MeSH Terms: conditions — Antithrombin III Deficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Citrated plasma Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antithrombin deficient patients: patients with proven, inherited antithrombin deficiency
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — No interventions planned: treatment of patients at the discretion of the treating/responsible physician

SUMMARY:
Inherited antithrombin deficiency is a rare autosomal dominant disorder that predisposes to the development of venous thromboembolism, even at young age.

Inherited AT deficiency is considered the most severe form of inherited thrombophilia, increasing up to 40 times the risk of venous thrombosis.

Our center has been performing research on antithrombin deficiency for several years. Therefore, it was decided to initiate a registry for patients with inherited antithrombin deficiency with the goal to gain more insight into what drives the development of a thrombotic event in patients with AT deficiency, both at the environmental level (lifestyle, management of risk situations, presence of additional thrombotic risk factors…) and at the genetic level.

DETAILED DESCRIPTION:
Background:

Antithrombin (AT) is the most important physiological inhibitor of blood coagulation, targeting predominantly factor X and thrombin (Factor II). It is a serine protease inhibitor encoded by the SERPINC1 gene and is synthesized in the liver. Inherited antithrombin deficiency is a rare autosomal dominant disorder that predisposes to the development of venous thromboembolism (VTE), even at young age. We can distinguish two types of AT deficiency: quantitative (type I) and qualitative (type II) deficiencies. According to which function of the protein is affected, type II deficiencies are subdivided into Heparin Binding Site (HBS), Reactive Site (RS) or Pleiotropic Effect (multiple functions or conformational consequences) deficiencies.

Inherited AT deficiency is considered the most severe form of inherited thrombophilia, increasing up to 40 times the risk of venous thrombosis. Antithrombin deficiency is a rare monogenic autosomal dominant disorder although the exact prevalence of AT deficiency remains largely unknown, probably because of the wide clinical heterogeneity. More than 400 different genetic variants in SERPINC1 have been identified. Diagnosis of AT deficiency is done by functional assays that are based on the inhibition of target proteases (Factor Xa or Factor IIa) in the presence of heparin. While biochemical, structural, and molecular information about AT is ample, there is a limited knowledge about the natural history of this disorder. The risk of venous thrombosis in carriers of AT deficiency is well documented but there are many important issues concerning the natural history of AT deficiency that must be unraveled: First, there is a remarkable heterogeneous presentation of AT deficiency. Type I deficiency has been associated with poorer prognosis than type II, but no systematic genotype-phenotype correlations have been done. Moreover, as for any other thrombotic disorder, we could expect that additional factors may modulate the risk of thrombosis in AT deficiency, even for carriers of the same genetic defect.

Objective In this study, the investigators will retrospectively and prospectively collect data on all AT deficient patients diagnosed in or referred to our center for diagnostic work up. The data will be used to create a national registry of antithrombin deficient patients.

The data collected in this registry will allow to gain more insight into what drives the development of a thrombotic event in patients with AT deficiency, both at the environmental level (lifestyle, management of risk situations, presence of additional thrombotic risk factors…) and at the genetic level. Data on obstetric complications and use of anticoagulant drugs will also be collected.

The study will help to assess the thromboembolic risk linked to distinct mutations and different (sub)types of AT deficiency. The findings could help steering the therapeutic attitude and give clinicians the opportunity to propose a more individually, patient-based approach for anticoagulation.

Furthermore, the observations will form the basis for more fundamental research into the pathophysiology of thrombosis in antithrombin deficient patients.

The registry will enroll as many confirmed or suspected hereditary AT deficiency patients as possible; there is no cap on enrollment. The registry enrollment and follow-up periods are open-ended. The endpoints for patients with confirmed or suspected hereditary AT deficiency are death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically confirmed antithrombin deficiency
* Patients with phenotypic antithrombin deficiency in which the genetic defect has not been elucidated yet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed inherited antithrombin deficiency are eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2060-12 (Estimated)

PRIMARY OUTCOMES:
Change in occurrence of thromboembolic events over time | Every 2 years for a period of 25 years or until death, whichever comes first
  Inquiry on occurrence of thromboembolic event by means of questionnaire
Change in occurrence of arterial thrombotic events over time | Every 2 years for a period of 25 years or until death, whichever comes first
  Inquiry on occurrence of arterial thrombotic event by means of questionnaire
Change in occurrence of obstetric complications over time | Every 2 years for a period of 25 years or until death, whichever comes first
  Inquiry on occurrence of obstetric complications by means of questionnaire

SECONDARY OUTCOMES:
Change in disease-modifying factors: thrombotic risk factors | Every 2 years for a period of 25 years or until death, whichever comes first
  collection of disease-modifying factors by means of questionnaire
Change in anticoagulant treatment | Every 2 years for a period of 25 years or until death, whichever comes first
  collect data on use of anticoagulant treatment by means of questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Orlando, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided